CLINICAL TRIAL: NCT02729441
Title: Perindopril vs Ramipril for Persistence in MAU Reduction Study
Acronym: ENDURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Servier (Industry)
Responsible Party: Principal Investigator, Sheldon Tobe, Staff Physician, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 053-2010
Record Dates: First submitted 2016-03-24; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Microalbuminuria
MeSH Terms: conditions — Diabetes Mellitus | interventions — Ramipril; Perindopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramipril (Active Comparator): Maximal recommended dose of ramipril "Altace®" (10 mg/d) given as an active comparator for 12 week.
  Interventions: Drug: ramipril
- Perindopril (Experimental): Perindopril "Coversyl®" at maximal recommended dose (8 mg/d) as experimental therapy for 12 weeks.
  Interventions: Drug: perindopril

INTERVENTIONS:
Drug: ramipril — Comparison of two renin angiotensin aldosterone inhibitors
  Other Names: Altace
  Arms: Ramipril
Drug: perindopril — Comparison of two renin angiotensin aldosterone inhibitors
  Other Names: Coversyl
  Arms: Perindopril

SUMMARY:
The investigators conducted a single center study controlled study involving 20 patients with Type 2 Diabetes and hypertension who were randomly assigned to receive ramipril 10mg or perindopril 8mg. The primary endpoint was difference in urine albumin-creatinine ratio at night time and during the day. Secondary endpoint was measurement of blood pressure.

DETAILED DESCRIPTION:
Design/Method This was a single arm, prospective, randomized, single blinded, open label cross-over study of the urine albumin excretion during the day and at night after 12 weeks of therapy with either perindopril 8 mg per day or ramipril 10 mg per day in people with diabetes. Men and women were eligible for the study if they met the following criteria: Age>18 years, type 2 diabetes with adequate blood sugar control (Hemoglobin A1c (A1c)<8.4%), therapy with ace inhibitor(ACEi) or angiotensin receptor blocker (ARB) for a period of 8 weeks prior to and throughout the screening period along with blood pressure (BP) <130/80 mmHg, known abnormal albuminuria for at least 12 weeks before screening and throughout the screening period as defined as (urine albumin by albumin-creatinine ratio (ACR) > 5.0 for men and women up to 50 mg/mmol).

Exclusion criteria included: women who were pregnant or lactating, women of childbearing age not on contraception, dual therapy with both ARB and ACEi, 8 weeks prior to screening visit or during screening period, allergy or history of cough with ACEi, known hypersensitivity to study medication diluent or to any constituent of study medication, poorly controlled hypertension (HTN) requiring a change of dose of ACEi or ARB within 8 weeks of screening visit, change in urine albumin by ≥ 2x from a previous level to the screening level while on stable drug dosing, myocardial infarction within 12 weeks of screening, congestive heart failure (NYHA Class IV), severe coronary artery disease, severe liver disease, renal artery stenosis.

Patients meeting the inclusion and exclusion criteria were enrolled in the study and randomized. Following this, eligible patients were switched from their existing renin angiotensin aldosterone system (RAAS) blocker to ramipril 10 mg daily for 1 week to determine if ramipril was tolerated. They then were entered into a stabilization phase of 12 weeks of uninterrupted ramipril therapy. Patients were assigned to receive either perindopril 8 mg once daily or 10 mg ramipril once daily based on the randomization code in an open label fashion. Treatment with either therapy was for 12 weeks each. At the end of these treatment periods patients were instructed to collect three sets of spot urine samples to reflect night and day urine albumin excretion. Additionally, patients were instructed to take four home blood pressure measurements, 2 in the morning and 2 in the evening. The morning recordings were to be done before the medication was taken. At the end of the 12 week treatment periods, measurements of urine electrolytes, A1c, urea, creatinine were also collected. A 24 hour ambulatory blood pressure monitoring (ABPM) was also completed at the end of the last two treatment periods.

Laboratory Procedures:

Ambulatory blood pressure was measured was performed over a period of 24 hours using a clinically validated device (model 90270, Spacelabs Medical Inc., Redmond, Washington, USA). The machine was instructed to measure blood pressure every 15 minutes throughout the day (7:00am to 11:00 PM) and every 30 minutes between 11:00pm and 7:00am. Patients were instructed to remain motionless every time the device was active. Values obtained were averaged each hour before calculating the day, night and average 24hr blood pressure.

During the 12th week of each treatment period, urine was collected from each patient to quantitatively measure urine sodium, potassium, urea, creatinine. AER was measured from urine collected under standard conditions. Three specimens were collected in each treatment period and the results were analyzed by immunoassay.

Statistical Analysis:

Statistical analysis of data was performed by means of SAS statistical software for Windows (SAS., Cary, North Carolina) with results being expressed as mean (SD).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes,
* stable therapy with an ACEi or ARB for 8 weeks prior to screening period
* blood pressure controlled to < 130/80 mmHg

Exclusion Criteria:

* Pregnancy,
* dual therapy with ACEi and ARB 8 weeks prior to screening
* history of cough with ACEi
* hypersensitivity to either medication
* myocardial infarction within 12 weeks of screening
* congestive heart failure (NYHA Class IV)
* severe coronary artery disease
* severe liver disease
* renal artery stenosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Urine albumin:creatinine ratio day and night | 24 hours
  spot urine samples
24 Hour Ambulatory Blood Pressure Monitoring | 24 hours
  24 hour, day, and night systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada